CLINICAL TRIAL: NCT00819923
Title: Comparison of Bio-Active-Stent to the Everolimus-Eluting Stent in Acute Coronary Syndrome (A Prospective, Randomized and a Multicenter Clinical Study)
Brief Title: Comparison of Bio-Active-Stent to the Everolimus-Eluting Stent in Acute Coronary Syndrome
Acronym: BASE-ACS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital District of Satakunta (Other)
Responsible Party: Pasi Karjalainen, MD, PhD, Department of cardiology, Satakunta Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SA-003
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Acute Coronary Syndrome
Keywords: Titanium; everolimus; drug eluting stent; stent thrombosis; restenosis; percutaneous coronary intervention; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients receiving bio-active stent during the intervention
  Interventions: Device: Percutaneous coronary intervention
- 2 (Active Comparator): Patients receiving everolimus-eluting stent during the intervention
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — Intra-coronary stenting
  Other Names: TITAN-2 stent,; Hexacath, France
  Arms: 1
Device: Percutaneous coronary intervention — Intra-coronary stenting
  Other Names: Promus (Boston,USA); Xience-V (abbott, Usa)
  Arms: 2

SUMMARY:
The purpose of the trial is to compare the safety and effectiveness of bio-active-stent (BAS) and everolimus-eluting stent (EES) in patients presenting with acute coronary syndrome.

DETAILED DESCRIPTION:
The BASE-ACS trial is an academic study, which will be conceived and conducted as a multicenter (multi-country) study by experienced interventional cardiologists. This study is independent of commercial interests.

The purpose of the trial is to compare the safety and effectiveness of bio-active-stent (Titan-2®) and everolimus-eluting stent (Xience V®, Promus®) in patients presenting with acute coronary syndrome.

A total of 850 patients will be included in the randomized study. The primary end point (MACE) is the composite of cardiac death, myocardial infarction and target lesion revascularization during 12 months of follow-up. Enrollment of patients will start in November 2008 and end in 2009.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting with acute coronary syndrome (unstable angina, non-st-elevation myocardial infarction or st-elevation myocardial infarction)and undergoing percutaneous coronary intervention
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* Expected survival < 1 year
* Allergy to aspirin, clopidogrel or ticlopidine
* Allergy to heparins, glycoprotein IIb/IIIa inhibitors or bivalirudin
* Allergy to everolimus
* Active bleeding or significant increased risk of bleeding
* Stent length longer than 28 mm needed
* Stent diameter > 4.0 mm needed
* Thrombolysis therapy
* Planned surgery within 12 months of PCI unless the dual antiplatelet therapy could be maintained throughout the perisurgical period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2008-11; Primary Completion 2013-05 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The primary end point (MACE) is the composite of cardiac death, myocardial infarction (MI) and target lesion revascularization (TLR) during 12 months of follow-up. | 12 months

SECONDARY OUTCOMES:
All cause death, cardiac death, MI, stent thrombosis and TLR at 1, 6, 12 and 18 months, and at 2, 3, 4 and 5 years. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pasi P Karjalainen, MD, PhD, Principal Investigator — Satakunta Central Hospital, Pori, Finland; Antti Ylitalo, MD, PhD, Principal Investigator — Satakunta Central Hospital, Pori, Finland; Matti Niemela, MD, PhD, Principal Investigator — Oulu University Hospital; Juhani KE Airaksinen, Professor, Principal Investigator — Turku University Hospital, Turku, Finland; Otto Hess, Professor, Principal Investigator — Bern University Hospital, Bern, Switzerland
Locations (6):
- Finland (6):
  - Helsinki University Hospital, Helsinki
  - Jyvaskyla Central Hospital, Jyväskylä
  - Keski-Pohjanmaan Keskusairaala, Kokkola
  - Oulu University Hospital, Oulu
  - Satakunta Central Hospital, Pori
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Karjalainen P, Kiviniemi TO, Lehtinen T, Nammas W, Ylitalo A, Saraste A, Mikkelsson J, Pietila M, Biancari F, Airaksinen JK. Neointimal coverage and vasodilator response to titanium-nitride-oxide-coated bioactive stents and everolimus-eluting stents in patients with acute coronary syndrome: insights from the BASE-ACS trial. Int J Cardiovasc Imaging. 2013 Dec;29(8):1693-703. doi: 10.1007/s10554-013-0285-8. Epub 2013 Aug 31. PMID 23996244